CLINICAL TRIAL: NCT05037253
Title: The Effect of Vitamin D Supplementation in Reducing COVID-19 Morbidity Among Healthcare Workers
Brief Title: COVID-19 Morbidity in Healthcare Workers and Vitamin D Supplementation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0811-20-01C
Record Dates: First submitted 2021-08-25; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: COVID-19 Respiratory Infection
Keywords: level of 25-hydroxyvitamin D; COVID-19 disease; Healthcare Workers
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Parallel Assigment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high dose (Active Comparator): Vitamin D therapy will initiate at a dosage of 50,000 IU on the first and second week, followed by a switch to a daily intake of 5,000 IU for 3 months.
  Interventions: Drug: Vitamin D
- Low dose: (Active Comparator): Vitamin D therapy will prescribe for 3 months at a dosage of 2,000 IU/day.
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Patients will be randomised to receive either high dose vitamin D (50,000 IU weekly) on the first and second week, followed by a switch to a daily intake of 5,000 IU for 3 months or low dose vitamin D (2,000 IU weekly) for 3 months.

SUMMARY:
[Aim] Purpose of the study: to analyze the effect of vitamin D supplementation in reducing COVID-19 morbidity and severity in healthcare workers.

The study will involve a minimum of 120 medical staff. All participants in the study will assess twice for serum 25(OH)D level: baseline and after 3 months of Vitamin D supplementation. After the baseline examination, the subjects will be randomized into 2 groups. In the first (No. 1), vitamin D therapy will initiate at a dosage of 50,000 IU on the first and second week, followed by a switch to a daily intake of 5,000 IU for 3 months. In the second group (No. 2), vitamin D therapy will prescribe for 3 months at a dosage of 2,000 IU/day. After 3 months of vitamin D supplementation, all participants will undergo to repeat testing of serum 25(OH)D level with an assessment of the effectiveness of the therapy. Body mass index (BMI), height, weight, SARS-CoV-2 antibodies (IgG), 25-hydroxycalciferol (25(OH)D) and presence of acute viral infection futures, parameters assessed after treatment.

DETAILED DESCRIPTION:
The COVID-19 pandemic that swept the world in 2019 radically changed not only the social sphere of life, subordinating everything around to its influence, but also the healthcare sector. It affected both its practical and scientific sides, globally changing the approach to medicine. Numerous studies around the globe are being conducted on the prevention and treatment of this infection. A significant amount of them study the role of vitamin D in the pathogenesis of the disease. Cholecalciferol (Vitamin D) is a fat-soluble vitamin that is involved in maintaining the serum calcium-phosphorus gradient. Vitamin D supplementation significantly reduces the risk of osteoporosis, and also affects the regulation of immune responses by modulating innate and adaptive immune responses. It has been shown to inhibit the proliferation of T cells, namely the subsequent transformation of Th1 cells to Th2 cells. This effect on cell proliferation and differentiation contributes to a significant decrease in the level of proinflammatory cytokines, thereby reducing the severity of immune-mediated damage. It was these mechanisms that formed the basis of the theory about the ability of vitamin D to prevent the severe course of coronavirus infection and even prevent it. At the moment, the effect of vitamin D on reducing COVID-19 morbidity is not fully confirmed.

Patients and Methods: Baseline characteristics will be recorded for all patients including medical history, height, weight, body mass index (BMI), antibodies to SARS-CoV-2 (IgG) and 25(OH)D. Serum 25(OH)D level, IgG to SARS-CoV-2 will be repeated at 12-14 weeks. Also, we will check information about clinical manifestation of COVID -19 and CT results in cases positive Ab. The research format is a prospective controlled single-center study. The study was carried out based on the Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health of the Russian Federation, October 30, 2020, to August 31, 2021. During the study, medical care workers who are working in an infectious hospital and who taking vitamin D in a controlled manner, having previously signed informed consent, will be observed. The study will be involved minimum 120 medical staff, including women and men. All subjects will be divided into three groups according to the criterion of having a higher, secondary, or no medical education. All participants in the study will be assessed twice for the level of 25-hydroxyvitamin D [25(OH)D], IgG to SARS-CoV-2 in their blood: before the start of therapy with cholecalciferol and after 3 months of Vitamin D administration. After the screening, the subjects will be randomized into 2 groups. In the Group 1, vitamin D therapy will be initiated at a dosage of 50,000 IU on the first and seventh week, followed by a switch to a daily intake of 5,000 IU for 12 weeks. In the Group 2, vitamin D therapy will be prescribed for 12 weeks at a dosage of 2,000 IU. After 3 months of taking vitamin D supplementation, all participants will undergo to repeat testing of the 25(OH)D level in the blood with an assessment of the effectiveness of the therapy. IgG titer and PCR results will be compared in two groups of participations taking different doses of vitamin D supplementation.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged 18 to 65 years
* who did not take Vitamin D supplementation
* healthcare workers, during the pandemic
* who had not previously tolerated new coronavirus infection

Exclusion Criteria:

* pregnancy or nursing
* a history of granulomatous diseases
* severe gastrointestinal diseases (clinically apparent malabsorption syndrome)
* liver disease
* kidney disease
* individual intolerance drug
* vitamin D supplementation
* drugs known to affect vitamin D metabolism (e.g., anticonvulsants, glucocorticoids, diuretics)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 antibodies (IgG) | [Baseline and 12 - 14 weeks
  COVID-19 presence in healthcare workers in infectious clinic will be determined by detection of IgG to SARS-CoV-2 (reference values: > 1.1 - positive test; < 0.8 - negative test; the result of 0.8 between 1.1 - boundary test) (Enzyme immunoassay kits - Vector-Best, Novosibirsk, Russia).
Positive PCR test | [Baseline and 12 - 14 weeks
  nasopharyngeal and oropharyngeal smear

SECONDARY OUTCOMES:
Serum 25(OH)D level | Baseline and 12 - 14 week
  Assessment the 25(OH)D level on different dose of Vitamin D supplementation and association between it's level with positive PCR and IgG levels
COVID-19 clinical features | Baseline and 12 - 14 week
  Fever, cough, myalgia, loss of smell or taste, abdominal pain, rhinorrhea and etc.
CT data | Baseline and 12 - 14 week
  Siemens Somatom Definition is a high-speed 128-slice CT scanner equipped with two X-ray tubes.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health of the Russian Federation, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No